CLINICAL TRIAL: NCT05760716
Title: The Effect of Prone Position Use on Ventilator Mode, Blood Gas and Ventilator-Associated Pneumonia in Intensive Care Patients
Brief Title: The Effect of Prone Position Use Ventilator-Associated Pneumonia in Intensive Care Patients
Acronym: prone
Status: Completed | Type: Observational
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Burcu DEDEOĞLU DEMİR, Assistant Professor, Istanbul Arel University
Other Study IDs: f8c2xi67
Record Dates: First submitted 2023-01-10; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Intensive Care Unit Syndrome
Keywords: prone position; Intensive care; ventilators mechanical; blood gas; ventilator- associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiment Group: * The prone position was positioned within the application steps.
  * The introductory characteristics form of the patients was filled in on the day the patient was included in the study.
  * Blood gas results and mechanical ventilator respiration indicators were followed up in the PP for 5-10 days and the changes were recorded in the tolerance hours.
  Arterial blood gas results, mechanical ventilator values, and ventilator-associated pneumonia status were monitored before the position was applied, during the position and after the patients were placed in the supine position by comparing the groups with and without the prone position.
  • Nursing intervention application steps for VAP were followed during the PP and the changes were recorded.
  Interventions: Other: practicing prone position
- Control Group: Routine nursing care was applied without any intervention. 'Patient Information Form', 'Patient Follow-up Charts', 'Clinical Pulmonary Infection Score', 'Braden Pressure Wound Risk Assessment' and 'Ramsey Sedation Scale' were used.

INTERVENTIONS:
Other: practicing prone position — Wash your hands. Prepare the materials. Before starting the procedure, inform the patient and explain the procedure. Ensure patient privacy. Raise the guardrail opposite the work area. Take the proper posture. Pay attention to body mechanics. Lay the patient on their back in the middle of the bed. Place a pillow under the patient's head to cover their shoulders. Extend arms to side of body with elbows slightly bent inward (flexion). Place a pillow under your arms. Place roller in palm. Place a thin pillow or a thinly folded towel/sheet under the waist. Place a thin towel under the knees. Support the bottom of the ankles with a pillow. Support the soles of the feet with a foot board. Raise the guardrail on the working side. Inform the patient that they can stay in this position for a maximum of 2 hours.
  Groups: Experiment Group

SUMMARY:
The aim of this experimental study was to investigate the effect of prone position use on ventilator values, blood gas and ventilator-associated pneumonia in intensive care unit patients. Between June 2021 and January 2022, 40 trials and 40 control patients were included in the intensive care units of two private hospitals and received mechanical ventilation support. The mechanical ventilator values, arterial blood gases and ventilator-related pneumonia conditions were evaluated and followed for at least 5 to 10 days just before the position was given by comparing the prone position (PP) and the patients were brought back into the supine position. The data were collected using 'Patient Follow-up Charts', 'Clinical Pulmonary Infection Score', 'Braden Pressure Half Risk Assessment' and 'Ramsey Sedation Scale' prepared in line with patient introduction form and evidence-based guidelines. In addition, life findings, cultural results and blood gas analyses were performed. Statistical analysis was performed using the 'NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah, USA)' program. 'Descriptive statistics, parametric and nonparametric tests' were used to evaluate the data. The level of statistical signiation was considered 'p<0.05'.

DETAILED DESCRIPTION:
Patients hospitalized in intensive care units are intubated and taken to mechanical ventilation support due to reasons such as inability to maintain airway patency, increase in respiratory/myocardial workload, and insufficient gas exchange. One of the strategies used to increase the effectiveness of mechanical ventilation therapy is the prone position (PP) application. In order to increase lung capacity and improve oxygenation in acute lung failure, the prone position was first applied in mechanical ventilation in the 1970s. Studies have shown that the prone position is protective against preventing ventilator-induced lung damage, and it has been found to increase PaO2/FiO2 in 70% of intensive care patients with severe hypoxemia receiving MV support. The reduction of the pressure on the lungs and the more homogeneous lung perfusion are effective in protecting the lungs in patients with prone position. Prone positioning of intensive care patients; It includes the risk of serious complications such as endotracheal tube obstruction, unplanned extubations, tachy and bradyarrhythmias, loss of venous and arterial access, cardiac arrest and pressure ulcer development in anterior body surface areas.

Positioning is one of the practices that nurses use by using their professional knowledge and skills. The positive effects of the position given to the patients in the intensive care unit on treatment and care are stated. Nurses continue to play a key role in the follow-up and treatment of patients who are placed in the prone position under mechanical ventilation therapy, from the continuous evaluation of the patients to the implementation of care practices, to provide the best clinical results.

In this study, a randomized controlled experiment was planned to determine the effect of the prone position by evaluating the mechanical ventilator values, blood gas and ventilator-associated pneumonia status before the position is applied, during the position and after the patients are brought back to the supine position by comparing the groups with and without the prone position.

The aims of the research;

* How prone position affects ventilator mode values
* How the prone position affects blood gas results,
* To examine how prone position affects the rate of development of ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Receiving respiratory support with a mechanical ventilator in the ICU,
* COVID 19 test negative,
* Consent by the first degree relative.

Exclusion Criteria:

* Being under the age of 18,
* Receiving a diagnosis of VAP before admission to the ICU,
* Having a positive COVID 19 test,
* Presence of an obstacle to prone positioning (obesity, pregnancy, anterior chest wall surgery, advanced heart failure, etc.).
* Not giving consent to participate in the study by a first-degree relative

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research was carried out between June and December 2021 in the 14-bed and 26-bed general intensive care units of two private hospitals on the European side of Istanbul.
  Power analysis was performed with the 'G*Power (v3.1.7) program' in the sample calculation. In general, studies should have 80% power. The power of the study is expressed as '1-β (β = II type error probability)'. Evaluations to be made with two independent groups; Since it is assumed to have a large effect size (d=0.8), according to the calculation made, it was determined that there should be at least 26 people in the groups at the level of 'α=0.05' according to Cohen's effect size coefficients. Considering that there may be losses during the study process, 40 people were included in each group.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | 3-5 minutes
  demographics
Patient Follow-up Charts | 15-20 minutes
  On vital signs

SECONDARY OUTCOMES:
Clinical Pulmonary Infection Score | 3-5 minutes
  'Clinical Pulmonary Infection Score' (CPES); It examines seven clinical parameters including leukocyte count, body temperature, endotracheal aspirate (ETA)/microbiological culture results, amount and character of tracheal secretion, Pa02/Fi02 ratio, and presence of pulmonary infiltration. A score of 6 or more suggests VIP.
Braden Pressure Sore Risk Assessment Scale | 5-8 minutes
  The 'Braden Pressure Sore Risk Assessment Scale' (BBIRRS) consists of '6 sub-dimensions' and '19 risk assessments'. 'Perception of stimulus, activity, movement, humidity, nutrition items are between 1-4 points; friction-tear is evaluated between 1-3 points. As the scores obtained from the scale decrease, the risk of developing pressure ulcers increases, individuals with a scale score of '3-14' are considered to be at 'moderate' risk for the development of pressure sores, and those with a score of '15-16' are considered to be 'low risk'. The total score of the scale varies between '6-23' points.
Ramsey Sedation Scale | 5-8 minutes
  The scale includes 1 to 6 points. 1 point: alert, anxious and/or restless, 2 points: alert, cooperative, oriented, calm, 3 points: sleeping, responding to verbal stimulus, 4 points: sleeping, moderately responding to painful stimulus , 5 points: sleeping, responding slowly to painful stimulus, 6 points: sleeping, no response to painful stimulus. The lowest score on the scale: 1: agitation, the highest score 6: deep sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Dedeoglu Demir B, Enc N, Borekci S. The effect of prone positioning on ventilator parameters, blood gas levels, and ventilator-associated pneumonia in intensive care unit patients: a randomized controlled trial. BMC Nurs. 2025 Feb 21;24(1):203. doi: 10.1186/s12912-025-02817-3. PMID 39984994